CLINICAL TRIAL: NCT02214537
Title: Embryo Development Measure Depending on the DNA Sperm Fragmentation
Brief Title: Does DNA Sperm Fragmentation Affects Embryo Morphokinetic?
Acronym: MACs-ESD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because we don´t have the necessary technology anymore
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, David Agudo Garcillan, PHD, IVI Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MADDA12201301
Record Dates: First submitted 2014-07-25; First posted 2014-08-12 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Blastocyst Time; Pronuclear Appearance; Pronuclear Fading; Embryo Compaction; Cleavage Times

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MACS (Experimental): Patients with MACS Selection
  Interventions: Other: MACS

INTERVENTIONS:
Other: MACS

SUMMARY:
The embryokinetics may be a new prognostic factor for choosing the human embryos with the highest implantation potential. In order to identify the factors that may affect the rate of embryo cleavage, there are many studies about morphokinetics and culture medium, oxygen tension, oocyte quality or type of medication used for ovarian stimulation. However there are no published data with respect to the influence of sperm DNA fragmentation in the embryo kinetic.

ELIGIBILITY:
Inclusion Criteria:

* Patients 36 to 38 years
* Fresh sample semen
* Minimum 6 oocytes
* Semen sample with at least 5 million/ml and at least 30% of progressive motile sperm.

Exclusion Criteria:

* Patients younger than 36 or older than 38 years old
* Frozen semen sample
* Less tan 6 oocytes.
* Semen samples with less than 5 million / ml or less than 30% of motile sperm.

Ages: 36 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Time of pronuclear appearance in hours. | The mean time of appearance of pronuclei is 3.3951 hours in our patients. We are going to evaluate pronuclear appearence time in hours in our study groups
  We want to study whether differences exist in the time of appearance of pronuclei in those embryos that derived from semen samples from the two study groups
  the minimum value of the difference to be detected; we said that about 3 hours apart.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Alonso, Study Director — IVI Madrid; David Agudo, PhD, Study Director — IVI Madrid; Maria Testillano, Study Chair — IVI Madrid; Alberto Pacheco, PhD, Study Director — IVI Madrid
Locations (1):
- IVI Madrid, Madrid, Spain